CLINICAL TRIAL: NCT05440773
Title: A Phase 2 Randomized, Controlled Study to Evaluate the Activity Level, Optimal Dosage, Safety, and Accepted Formulation of Artemisia Afra Tea Infusions in Eliminating Plasmodium Reservoirs in Malaria Endemic Areas of Cameroon and Rwanda
Brief Title: Emptying Malaria Reservoirs to Accelerate Malaria Elimination in High Transmission Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xxxxx
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Asymptomatic Malaria
Keywords: Artemisia infusions, Plasmodium reservoirs, malaria endemic areas

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment group 1 (TG 1) (Experimental): Group of 8 persons receiving A. afra infusions of 5g/1liter of water, 3drinks a day, daily for 1week (7 days) (current recommendation)
  Interventions: Other: Artemisia afra tea infusions
- Treatment group 2 (TG 2) (Experimental): Group of 8 persons receiving A. afra infusions of 5g/500ml of water, 2drinks a day, daily for 1week (7 days) (increase concentration and decrease dose frequency).
  Interventions: Other: Artemisia afra tea infusions
- Treatment group 3 (TG 3) (Experimental): Group of 8 persons receiving A. afra infusions,5g/1liter of water, 3drinkss a day, weekly for 4weeks (decrease dose frequency and increase length of treatment).
  Interventions: Other: Artemisia afra tea infusions
- Treatment group 4 (TG 4) (Experimental): Group of 8 persons receiving flavored A. afra infusions, 5g/1liter of water, 3drinks a day, daily for1week (7 days) (current treatment with improved taste).
  Interventions: Other: Artemisia afra tea infusions
- Treatment group 5 (TG 5) (Experimental): Group of 8 persons flavored A. afra infusions, 5g/500ml of water, 2drinks a day, daily for 1 week (7 days) (improved taste, increase concentration and decrease dose frequency).
  Interventions: Other: Artemisia afra tea infusions
- Treatment group 6 (TG 6) (Experimental): Group of 8 persons receiving flavored A. afra infusions, 5g/1liter of water, 3drinks a day, weekly for 4weeks (improved taste, decrease dose frequency and increase length of treatment).
  Interventions: Other: Artemisia afra tea infusions
- Treatment group 7 (Placebo Comparator): Group of 4 persons receiving flavored placebo infusions, 5g/liter of water, 3drinks a day, daily for 1week (7 days) (improved taste with no active molecule)
  Interventions: Other: Flavored placebo infusions
- Treatment group 8 (Placebo Comparator): Group of 4 participants receiving regular tea placebo taken as desired, daily for 1 week (7 days) (Regular tea with no active molecule).
  Interventions: Other: Regular tea placebo

INTERVENTIONS:
Other: Artemisia afra tea infusions — A. afra infusions of 5g/1litter of water, 3drinks a day, daily for 1week (7 days) (current recommendation).
  Arms: Treatment group 1 (TG 1)
Other: Artemisia afra tea infusions — A. afra infusions of 5g/500ml of water, 2drinks a day, daily for 1week (7 days) (increase concentration and decrease dose frequency).
  Arms: Treatment group 2 (TG 2)
Other: Artemisia afra tea infusions — A. afra infusions,5g/1liter of water, 3drinkss a day, weekly for 4weeks (decrease dose frequency and increase length of treatment).
  Arms: Treatment group 3 (TG 3)
Other: Artemisia afra tea infusions — A. afra infusions, 5g/1liter of water, 3drinks a day, daily for1week (7 days) (current treatment with improved taste).
  Arms: Treatment group 4 (TG 4)
Other: Artemisia afra tea infusions — A. afra infusions, 5g/500ml of water, 2drinks a day, daily for 1 week (7 days) (improved taste, increase concentration and decrease dose frequency).
  Arms: Treatment group 5 (TG 5)
Other: Artemisia afra tea infusions — Group of 8 persons receiving flavored A. afra infusions, 5g/1liter of water, 3drinks a day, weekly for 4weeks (improved taste, decrease dose frequency and increase length of treatment).
  Arms: Treatment group 6 (TG 6)
Other: Flavored placebo infusions — Flavored placebo infusions, 5g/liter of water, 3drinks a day, daily for 1week (7 days) (improved taste with no active molecule)
  Arms: Treatment group 7
Other: Regular tea placebo — Regular tea placebo taken as desired, daily for 1 week (7 days) (Regular tea with no active molecule).
  Arms: Treatment group 8

SUMMARY:
The study is a Phase 2 randomized controlled, partial-blind, parallel group study in plasmodium infected asymptomatic adults 18 years and older, with 8 study arms. It will use the adapted Zelen design, which has two steps in the consent process. In the first step, there is an informed consent from all participants for a cohort lifestyle study. According to this consent, participants are randomized without knowledge about the detailed protocol.

In the second step, only participants from the intervention group will receive the information about the intervention and the second consent will be obtained from them. The participants who will decline to participate to an intervention will continue in the cohort study, as the control group.

DETAILED DESCRIPTION:
This study will use the adapted Zelen design which has two steps in the consent process. At step one, informed individuals (students and workers) will be invited to participate in a screening and cohort survey on asymptomatic malaria, aimed at understanding the comportment of plasmodium parasite in asymptomatic plasmodium carriers over time. After informed consent is obtained during the first encounter (day 0), baseline assessments will be done and sociodemographic variables, clinical/medical history, physical assessment, prior medications information and participants' contact details will be recorded. Blood samples will be collected from each participant and examined for the presence of parasites (Gametocytes) using malaria rapid diagnostic test kit (mRDT). RDT positive samples will be re-examined with qPCR (quantitative polymerase chain reaction) and direct microscopy for confirmation. The qCPR will be repeated for negative samples and participants excluded if still negative. All qPCR positive samples will be further analyzed with rt PCR (real time polymerase chain reaction), for parasite quantification and specific stage identification, targeting specific parts of the gametocyte genes. Participants who fulfil the inclusion criteria will be randomly allocated in the 8 study arms in a 2:2:2: 2:2:2:1:1 ratio for the 6 treatment and 2 control arms, respectively. In the second step, only participants from the intervention groups will receive the information about the intervention and a second consent will be obtained from them (TG1-TG7). Treatment administration will be based on the allocation arm. The treatments will consist of Artemisia afra tea infusions for the 6 trial arms versus flavored placebo infusions and desired regular tea for the 2 control arms. The participants who will decline to participate to an intervention will continue in the cohort study, as a control group on regular tea (TG 8).

During 4 consecutive weeks, all participants will be tested using rtPCR once a week on Day 7, 14, 28 and 35, in order to assess gametocyte elimination rate with teas. During the 4 weeks, participants will be monitored and encouraged to comply to the prescribed treatment, and also monitored/assessed for any clinical symptoms and treatment reactions (ASEs and AE).

ELIGIBILITY:
Inclusion Criteria:

* Be student or worker of a participating University.
* Be 18 years and above, and in good general health condition.
* Have a device (phone, tablet, etc) that will support remote visits.
* Sign written informed consent form.
* Screened positive for malaria (RDT + and qPCR +) but asymptomatic.

Exclusion Criteria:

* To have a known hypersensitivity to any ingredients of the tea.
* Currently taking a malaria drug for prevention or treatment.
* To have participated in another malaria drug trial or device in the last 14days.
* To have a history or presence of clinically significant medical, psychiatric, or emotional condition.
* Reported diabetic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Decrease in parasite load over time | 4 weeks

SECONDARY OUTCOMES:
Decrease in gametocyte load in carriers with Artemisia afra tea by dose concentration, dose frequency, length of treatment, and formulation. | 4weeks
Acceptability (adherence and completion) of Artemisia afra treatment by dose concentration, dose frequency, length of treatment, and formulation (flavor). | 4weeks
Safety (ASEs) of Artemisia afra treatment in participants by dose concentration, dose frequency length of treatment, and treatment formulation. | 4weeks
Likelihood and variability in the rate of reservoir elimination with treatment, compliance/ acceptability, and occurrence of side effects /adverse events in different treatment arms. | 4weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suh Nchang Abenwie, MSc. MPH, Principal Investigator — UCLouvain, Bruxells -Belgium; Robert Annie, Professor, Study Director — Université Catholique de Louvain; Souopgui Jacob, Professor, Study Chair — Université Libre de Bruxelles; Ghogomu Stephen, Professor, Study Chair — University of Buea, Cameroon; Frederick Michel, Professor, Study Chair — Université de Liège

IPD SHARING:
Plan to Share IPD: No
No plan available.